CLINICAL TRIAL: NCT06837389
Title: Early Clinical Study of JY306 Universal NK Cell Injection in the Treatment of Adult Relapsed or Refractory CD70+ Malignant Hematologic Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-1013
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Relapsed or Refractory Hematological Malignancies
MeSH Terms: conditions — Recurrence; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JY306 universal NK cell injection (Experimental)
  Interventions: Biological: JY306 universal NK cell injection

INTERVENTIONS:
Biological: JY306 universal NK cell injection — "3+3" dose escalation trial

SUMMARY:
1. Primary objectives of study:To valuate the tolerability and safety of JY306 in patients with relapsed or refractory CD70 + malignant hematological tumors.
2. Secondary objectives of study:To conduct a preliminary Evaluation of the Efficacy, Pharmacokinetics, and Pharmacodynamics of JY306 in Patients with Relapsed or Refractory CD70+ Malignant Hematological Tumors.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory malignant hematological tumors judged by clinical diagnosis;
* The tumor cells were confirmed positive for CD70 by flow cytometry (FCM) or immunohistochemistry, and the positivity rate was >80%;
* Age 18-75 years (inclusive);
* The expected survival period from the signing date of the informed consent is more than 3 months;
* KPS≥80 points;
* The function of vital organs needs to meet the following conditions: 1) EF >50%, and there is no obvious abnormality in ECG; 2)SpO2≥90%; 3) Cr≤2.5ULN;4) ALT and AST≤5ULN, TBil≤3ULN;
* Subjects with pregnancy plans must agree to use contraception prior to enrollment in the study and after six months of study duration; If the subject is pregnant or suspects pregnancy, the investigator should be notified immediately;
* The subject or guardian understands and signs the informed consent form;

Exclusion Criteria:

* Have a New York Heart Association (NYHA) classification ≥III heart failure or myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically prominent heart disease within one year prior to signing the informed consent form, Or QTc interval >480ms (QTc interval is calculated by Fridericia formula) during screening;
* Those who have active GvHD, or need to use immunosuppressants;
* Have been diagnosed with malignant tumors other than primary tumors within 5 years prior to screening, except for adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ of the breast after radical resection;
* There are active infections or uncontrollable infections that require systemic treatment (excluding mild urinary and genital tract infections and upper respiratory tract infections) within 7 days prior to screening;
* History of autoimmune diseases (such as rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease) requiring systemic immunosuppressive/systemic disease-modifying drugs within the past 2 years;
* At screening, those with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HbcAb), and peripheral blood hepatitis B virus (HBV) DNA levels above the lower limit of detection; those with positive hepatitis C virus (HCV) antibody and positive peripheral blood HCV RNA; those with positive human immunodeficiency virus (HIV) antibody; those with positive cytomegalovirus (CMV) DNA; those with positive Epstein-Barr virus (EBV) DNA; and those with positive Treponema pallidum particle agglutination (TPPA) test for syphilis should all be excluded;
* Subjects who have participated in other clinical trials within 4 weeks prior to signing the informed consent form, or for whom the date of signing the informed consent form is still within 5 half-lives of the last dose of the drug from the previous clinical trial (whichever is longer).
* Have a history of severe allergy to biological products;
* Unstable systemic diseases judged by the investigator: including but not limited to severe hepatic, renal or metabolic diseases requiring drug treatment;
* Pregnant or lactating women, and female subjects who plan to become pregnant within 2 years after cell infusion or male subjects whose partners plan to become pregnant within 2 years after cell infusion;
* According to the judgment of the investigator conditions that may increase the subject's risk or interfere with the trial results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence frequency, number of cases, incidence rate and severity of adverse events and adverse reactions occurring after infusion and before withdrawal or the safety follow-up period | From enrollment to one year after infusion